CLINICAL TRIAL: NCT03048968
Title: The Effect of a Walking Assist Robot on Gait Function and Brain Activity in Stroke Patients and Elderly Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: Samsung Electronics (Industry)
Responsible Party: Principal Investigator, Yun-Hee Kim, Professor, MD, PhD, Samsung Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2016-07-093
Record Dates: First submitted 2017-02-06; First posted 2017-02-09 (Estimated); Last update posted 2019-04-29 (Actual); Status verified 2019-04

CONDITIONS: Stroke; Healthy
Keywords: Exoskeleton Device; elderly; stroke
MeSH Terms: conditions — Stroke | interventions — Gait; Stair Climbing; Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group1: elderly adults (Experimental): Gait, sit-to-stand movement, stair climbing and treadmill gait with GEMS and without GEMS
  Interventions: Procedure: Gait, sit-to-stand movement, stair climbing and treadmill gait; Device: gait enhancing mechatronic system (GEMS); Device: treadmill
- study group2: stroke patients (Experimental): Sit-to-stand movement and treadmill gait with GEMS and without GEMS
  Interventions: Procedure: Sit-to-stand movement and treadmill gait; Device: gait enhancing mechatronic system (GEMS); Device: treadmill

INTERVENTIONS:
Procedure: Gait, sit-to-stand movement, stair climbing and treadmill gait — Spatio temporal characteristics, muscle activation and foot pressure distribution are measured by motion capture system, surface electromyography (sEMG) and F-Scan Mobile system during 10m walking test. Muscle activation and foot pressure distribution are measured by surface electromyography (sEMG) and F-Scan Mobile system during five times sit-to-stand test.Muscle activation and foot pressure distribution are measured by surface electromyography (sEMG) and F-Scan Mobile system during stair climbing. Cortical activation is measured by functional Near-Infrared-Spectroscopy (fNIRS) (NIRScout, NIRx, Germany) during treadmill gait.
  Arms: study group1: elderly adults
Procedure: Sit-to-stand movement and treadmill gait — Muscle activation and foot pressure distribution are measured by surface electromyography (sEMG) and F-Scan Mobile system during five times sit-to-stand test. Cortical activation is measured by functional Near-Infrared-Spectroscopy (fNIRS) (NIRScout, NIRx, Germany) during treadmill gait.
  Arms: study group2: stroke patients
Device: gait enhancing mechatronic system (GEMS) — Gait, sit-to-stand movement, stair climbing and treadmill gait with GEMS and without GEMS in elderly adults.
  Sit-to-stand movement and treadmill gait with GEMS and without GEMS in stroke patients.
Device: treadmill — Cortical activation is measured by functional Near-Infrared-Spectroscopy (fNIRS) (NIRScout, NIRx, Germany) during treadmill gait.

SUMMARY:
The purpose of this study was to investigate the effects of the new wearable hip assist robot, gait enhancing and motivating system (GEMS) developed by Samsung Advanced Institute of Technology (Samsung Electronics Co, Ltd., Korea) on gait, sit-to-stand movement and cortical activation in elderly adults and stroke patients.

DETAILED DESCRIPTION:
In elderly adults,

1. Spatio temporal characteristics, muscle activation and foot pressure distribution are measured by motion capture system (Motion Analysis Corporation, Santa Rosa, CA, USA), surface electromyography (sEMG) (Noraxon Inc., Scottsdale, AZ, USA) and F-Scan Mobile system (Tekscan Inc., South Boston, MA, USA) during 10m walking test.
2. Muscle activation and foot pressure distribution are measured by surface electromyography (sEMG) and F-Scan Mobile system during five times sit-to-stand test.
3. Muscle activation and foot pressure distribution are measured by surface electromyography (sEMG) and F-Scan Mobile system during stair climbing.
4. Cortical activation is measured by functional Near-Infrared-Spectroscopy (fNIRS) (NIRScout, NIRx, Germany) during treadmill gait.

In stroke patients,

1. Muscle activation and foot pressure distribution are measured by surface electromyography (sEMG) and F-Scan Mobile system during five times sit-to-stand test.
2. Cortical activation is measured by functional Near-Infrared-Spectroscopy (fNIRS) (NIRScout, NIRx, Germany) during treadmill gait.

ELIGIBILITY:
Inclusion Criteria:

* Elderly adults

  1. Age: between 65 and 84 years
  2. elderly adults who had no neurological or musculoskeletal abnormalities affecting gait
  3. Ability to walk at least 10m regardless of assist devices
* Stroke

  1. Age: between 20 and 84 years
  2. ≥ 3 months post stroke
  3. Ability to walk at least 10m regardless of assist devices
  4. Adequate gait function (FAC > 3)
  5. Physician approval for patient participation

Exclusion Criteria:

* Elderly adults

  1. History of any diseases (eg. lower extremity orthopedic diseases, neurologic disorders, cardiovascular disease, heart failure, uncontrolled hypertension that affect walking capacity, efficiency, and endurance)
  2. Severe visual impairment or dizziness that increases the risk of falls
* Stroke

  1. Serious cardiac conditions (hospitalization for myocardial infarction or heart surgery within 3 months, history of congestive heart failure, documented serious and unstable cardiac arrhythmias, hypertrophic cardiomyopathy, severe aortic stenosis, angina or dyspnea at rest or during activities of daily living)
  2. Advanced liver, kidney, cardiac, or pulmonary disease
  3. History of concussion in last 6 months
  4. History of unexplained, recurring headaches, epilepsy/seizures/skull fractures or skull deficits
  5. Preexisting neurological disorders such as Parkinson's disease, Amyotrophic Lateral Sclerosis (ALS), Multiple Sclerosis (MS), dementia

Ages: 20 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-10-23 (Actual)

PRIMARY OUTCOMES:
Cortical activation | 30minutes
  Cortical activation is measured by functional Near-Infrared-Spectroscopy (fNIRS) (NIRScout, NIRx, Germany) during treadmill gait.

SECONDARY OUTCOMES:
Berg Balance Scale (BBS) | 30minutes
  The BBS is a 14-item objective measure designed to assess static balance and fall risk in adult populations and is a well-accepted measure in the stroke literature. The functional activities that are assessed include sitting and standing balance during transfers, altered base of support, reaching, turning, eyes open and closed.
Fall Efficacy Scale (FES) | 20minutes
  Fall Efficacy Scale (FES) is a 10-item questionnaire designed confidence in their ability to perform 10 daily tasks without falling as an indicator of how one's fear of falling impacts physical performance. Each item is rated from 1 ("very confident") to 10 ("not confident at all"), and the per item ratings are added to generate a summary total score.
Manual Muscle Test (MMT) | 20minutes
  Manual muscle testing (MMT) is a procedure for the evaluation of the function and strength of individual muscles and muscle groups based on the effective performance of a movement in relation to the forces of gravity and manual resistance.
Range of Motion (ROM) | 20minutes
  Range of Motion (ROM) testing is the measurement of movement around a specific joint or body part.
Functional Ambulation Classification (FAC) | 20minutes
  The Functional Ambulation Categories (FAC) is a functional walking test that evaluates ambulation ability. This 6-point scale assesses ambulation status by determining how much human support the patient requires when walking, regardless of whether or not they use a personal assistive device.
The modified Rankin Scale (mRS) | 20minutes
  The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability.
Change in 10 meter walk test from baseline in gait speed | 1hour
  Measure of self selected speeds by measuring the time it takes an individual to walk 10 meters. To perform the test, patient walks 10 meters (33 ft) and the time is measured when the leading foot crosses the start line and the finish line. The instructions are: "Please walk this distance at your normal pace when I say go."

CONTACTS AND LOCATIONS:
Overall Officials: Yun-Hee Kim, Study Chair — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee SH, Lee HJ, Shim Y, Chang WH, Choi BO, Ryu GH, Kim YH. Wearable hip-assist robot modulates cortical activation during gait in stroke patients: a functional near-infrared spectroscopy study. J Neuroeng Rehabil. 2020 Oct 29;17(1):145. doi: 10.1186/s12984-020-00777-0. PMID 33121535